CLINICAL TRIAL: NCT02930681
Title: Double-blind, Randomised, Placebo-controlled, 3-way Cross-over Study to Evaluate the Benefit of Two Glucosanol™ Dosages to Reduce Post-prandial Glucose Levels in Overweight Subjects
Brief Title: Efficacy of Glucosanol™ in Reducing Post-prandial Glucose Levels in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INQ/024515
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Hyperglycemia, Postprandial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Four capsules of placebo to be taken 30 mins before each test meal at the investigator's site
  Interventions: Dietary Supplement: Placebo
- Glucosanol 1000mg (Experimental): Two capsules of placebo and two capsules of Glucosanol 500mg capsules to be taken 30 mins before each test meal at the investigator's site
  Interventions: Dietary Supplement: Glucosanol 500mg; Dietary Supplement: Placebo
- Glucosanol 2000mg (Experimental): Four capsules of Glucosanol 500mg to be taken 30 mins before each test meal at the investigator's site
  Interventions: Dietary Supplement: Glucosanol 500mg

INTERVENTIONS:
Dietary Supplement: Glucosanol 500mg
  Arms: Glucosanol 1000mg; Glucosanol 2000mg
Dietary Supplement: Placebo
  Arms: Glucosanol 1000mg; Placebo

SUMMARY:
Glucosanol had previously been proven to be effective in aiding weight loss and weight loss maintenance. Studies have also shown that Glucosanol (also known as Phaseolamin), was effective in aiding weight loss and also has evidence on reducing post-prandial glucose levels. This study is to enrich the existing evidence on dose-dependent post-prandial glucose effects of Glucosanol

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males and females, 18 to 65 years old
* Body mass index (BMI) 25.0-29.9 kg/m2
* Generally in good health
* Normal fasting blood glucose (FBG) 3.9- <5.6 mmol/L (70- <100 mg/dL) and glycated hemoglobin HbA1c of 4- <5.7 %
* Readiness to adhere to consumption of test meals and defined restrictions prior to test meals (refer to section 11.8 for details)
* Readiness to adhere to habitual lifestyle during the study, in particular to:

  1. maintain the same level of physical activity during the study, including non-strenuous transportation to the study visits
  2. if smoking, regular smoking at the same level as prior
* to the study and no smoking on days of test meals
* prior and during the visit
* Stable body weight in the last 3 months prior to V1 (≤5% self-reported change)
* Stable concomitant medications (if any) for at least last 3 months prior to V1
* Women of child-bearing potential only:

  1. negative pregnancy testing (ß-HCG in urine at V1)
  2. commitment to use reliable contraception methods

Exclusion Criteria:

* Known sensitivity to any ingredients / excipients of the IP
* Known food allergy (e.g. to cow's milk, eggs, wheat, crustacean, nuts etc.)
* Clinically relevant excursions of safety parameters
* Digestion/absorption disorders in gastrointestinal (GI) tract (e.g. inflammatory bowel disease)
* Uncontrolled hypertension >140/90 mmHg at V1
* Uncontrolled thyroid disorder at V1
* Any serious condition or disease that renders subjects ineligible
* Change in daily dose of any treatment and/or use of supplements with a possible impact on glycemic control in the last 3 months prior to V1 and throughout the study (refer to section 10 for details)
* Use of any anti-diabetic treatment or use of treatment and/or supplementation, for reduction of blood glucose levels within the last 4 weeks before V1 and throughout the study
* Use of medications or dietary supplements that may influence body weight ≤4 weeks and gastrointestinal functions ≤2 weeks prior to V1 and during the study
* Antibiotic and cortisone therapy ≤2 weeks prior to V1 and during the study
* Vegetarians and subjects with self-reported diet high in fat or protein
* Strenuous exercise within one day prior to each blood glucose sampling (including V1)
* History of bariatric surgery, small bowel resection or extensive bowel resection
* Recent blood donation within ≤1 month prior to study
* Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits) and any alcohol consumption within 24 h before blood glucose sampling
* Inability to comply with study procedures
* Pregnancy or nursing
* Participation in another study during the last 30 days of the screening visit (V1)
* Any other reason deemed suitable for exclusion, per investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in total PPG between verum 1000mg and 2000mg study arms vs the placebo study arm | 120 mins
  Change defined as incremental AUC0 - AUC120min in mmol/(L*min)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No